CLINICAL TRIAL: NCT01386034
Title: Effects of Oral Citrulline on Protein Metabolism in Patients With Intestinal Failure : a Prospective, Randomized, Double-blind, Cross-over Study
Brief Title: Effects of Oral Citrulline on Protein Metabolism in Patients With Intestinal Failure (Citrugrêle 2)
Acronym: CITRUGRELE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BRD/09/05-W
Record Dates: First submitted 2011-06-24; First posted 2011-06-30 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2016-05

CONDITIONS: Intestinal Failure
Keywords: Nutrition, protein metabolism, stable isotopes, mass spectrometry, intestinal failure
MeSH Terms: conditions — Intestinal Failure | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Citrulline/Placebo (Experimental)
  Interventions: Drug: Citrulline and placebo
- Placebo/Citrulline (Experimental)
  Interventions: Drug: Citrulline and placebo

INTERVENTIONS:
Drug: Citrulline and placebo — After receiving a 7-day oral supplementation with either citrulline or placebo, each subject will be admitted for a half day, after an overnight fast, and will receive a 5-h intravenous infusion of L-[1-13C]leucine. At regular intervals throughout the isotope infusion, blood will be obtained to measure 13C-enrichment in plasma a-keto-isocaproate, using gas chromatography-mass spectrometry. Simultaneously, 13C-enrichment will be measured in aliquots of expired air CO2 using isotope ratio mass spectrometry, and total CO2 production (VCO2) will be measured using direct calorimetry, respectively. Then the subject take no treatment for 13 days. The study will then be repeated a second time in an identical fashion, after a second 7-day period of oral supplementation with either citrulline or placebo.

SUMMARY:
The specific aim of this study is to determine whether oral citrulline administration enhances whole body protein synthesis in patients with intestinal failure. Protein metabolism will be assessed using an intravenous infusion of stable isotope labeled leucine. The investigators hypothesize that citrulline supplementation will decrease leucine oxidation without altering proteolysis, and consequently stimulate protein synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Adult between 18 and 75 years
* Patient with short bowel syndrome
* Patient with an incompetent small intestine after intestinal resection
* Patient fed orally and beyond more than 6 weeks after surgery
* Absence of any earlier supplementation with citrulline, glutamine, ornithine a-ketoglutarate, or stimol®
* No current artificial feeding (parenteral)
* No low-sodium diet- No renal, cardiac, respiratory or hepatic insufficiency
* No chronic inflammatory disease (intestinal or other)
* No current corticosteroid treatment
* Fasting blood glucose below 6mmol/L
* Patient able to understand benefits and risks of protocol
* Women who are of childbearing potential must have a negative serum pregnancy test and agree to use a medically acceptable method of contraception throughout the study and for 15 days following the end of the study
* Signed informed consent

Exclusion Criteria:

* Subject not fulfilling inclusion criteria
* Subject mentioned in articles L1121-5 to L1121-8 of "code de la santé publique"
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
whole body protein synthesis
  To determine whether oral citrulline administration enhances whole body protein synthesis in patients with intestinal insufficiency, as measured using an intravenous infusion of stable isotope labelled leucine.

SECONDARY OUTCOMES:
nitrogen balance
  Using a 6-h urine collection, to determine the effect of oral citrulline administration on nitrogen balance
Measure of insulin
  to determine whether the putative protein anabolic effect of citrulline is mediated by insulin or insulin-like-growth factor 1 (IGF-1), based on measurement of their plasma concentrations
Measure of insulin-like-growth factor 1 (IGF-1)
  To determine whether the putative protein anabolic effect of citrulline is mediated by insulin or insulin-like-growth factor 1 (IGF-1), based on measurement of their plasma concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique DARMAUN, Pr, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - Nantes University Hospital, Nantes
  - Clinique Saint Yves, Rennes

REFERENCES:
- [Derived] Jirka A, Layec S, Picot D, Bernon-Ferreira S, Grasset N, Flet L, Thibault R, Darmaun D. Effect of oral citrulline supplementation on whole body protein metabolism in adult patients with short bowel syndrome: A pilot, randomized, double-blind, cross-over study. Clin Nutr. 2019 Dec;38(6):2599-2606. doi: 10.1016/j.clnu.2018.12.030. Epub 2019 Jan 2. PMID 30642738